CLINICAL TRIAL: NCT06067373
Title: Impact and Burden of Postponing Elective Surgeries in Patients With Urological Diseases
Brief Title: Impact and Burden of Postponing Elective Surgeries
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 35-322 ex 22/23
Record Dates: First submitted 2023-08-28; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Mental Impairment; Complication
Keywords: postponed surgery
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with postponed surgery: patients with postponed surgery
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — After agreeing to participate, the patients receive a questionnaire in paper form.
  This consists of a total of 12 higher-level self-compiled questions as well validated survey instruments. The free questions relate, among other things, to to the surgery postponement, the associated burden, complications occurred, Effects on the employment situation, as well as the current state. The following validated survey instruments are used in the questionnaire: the NCCN Distress Thermometer to record the mental stress, a Severity Symptom Scale to record the symptom burden and the PROMIS-10 for recording the health-related life quality.

SUMMARY:
Overall, little is known about the effects and burdens of postponed operations in patients with urological diseases. To investigate the consequences and develop possible strategies for overcoming these challenges, the investigators would like to evaluate the influence of operation shifts in more detail.

DETAILED DESCRIPTION:
Medical care in Austria is struggling with staff shortages and consecutive OR (operating room) closures. The current development seems to be the result of problems that have been postponed for a long time to be accelerated by the COVID-19 pandemic. The introduction of COVID-19 vaccination and the establishment of protective measures and handling standards with infected patients made it possible to return to the regular operation. However, there is currently no noticeable improvement in the overall situation. The increasing shortage of nursing care in Austria is an increasingly urgent reason for this that affects all hospitals and care facilities. By prioritizing oncological interventions and an "oncology first" strategy at least oncological interventions and emergency interventions are performed on time. However, just looking at the waiting times for oncological interventions does not provide sufficient information of the current overall situation. The impairment for Patients with non-oncological diseases have received little attention so far given. Postponing elective surgery in patients with functional urological diseases (e.g. benign prostatic hyperplasia) can have a long-term impact on patient health and also means shifting their Surgery Burden and the stress for the patient. An American Study observed a decrease in prostate cancer diagnoses and an increase in diagnostic delays and postponements of treatments due to the pandemic, which led to greater stress and uncertainty in the affected patients.

The primary goal of this study is to record the burden on patients caused by the postponement of their surgery (mentally, physically).

Secondary outcomes include complication rates from postponement of surgery, effects on employment, awareness of the current situation (lack of care), state of health of patients upon admission to elective surgery.

ELIGIBILITY:
Inclusion Criteria:

- All patients over the age of 18 attending the Department of Urology for an elective surgery

Exclusion Criteria:

* lack of ability to give consent
* emergency operations

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the Urology department for elective surgery are eligible for the study and, if interested, receive the patient information.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
physical burden caused by postponement of elective surgery | depending on the interval of the postponed surgery; through study completion, an average of 1 year
  to evaluate the physical burden (e.g., scale 1-5 on severity of disease burden) caused by postponement of elective surgery
mental burden caused by postponement of elective surgery | depending on the interval of the postponed surgery; through study completion, an average of 1 year
  to evaluate the mental burden (e.g., scale: NCCN-Distress thermometer, scale 1-10) caused by postponement of elective surgery

SECONDARY OUTCOMES:
complication rates | depending on the interval of the postponed surgery; through study completion, an average of 1 year
  to evaluate the frequency complications (e.g., questions on urinary retention, comparison to patient records) caused by postponement of elective surgery
effect on employment | depending on the interval of the postponed surgery; through study completion, an average of 1 year
  to evaluate the effect on employment (e.g., questions about incapability to work, days of work leave, risk of getting unemployed) caused by postponement of elective surgery
awareness of the current situation | depending on the interval of the postponed surgery; through study completion, an average of 1 year
  to evaluate the awareness of the current situation (e.g, knowledge about the current situation of lack of personnel and resources)
general health status | depending on the interval of the postponed surgery; through study completion, an average of 1 year
  to evaluate global health status via PROMIS-10 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Medical University Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No